CLINICAL TRIAL: NCT06760728
Title: Multicenter Observational Study on the Prevalence of Inappropriate Prescribing in Elderly Patients At Admission and Discharge from a Hospital Ward Using the STOPP/START Criteria
Brief Title: Inappropriate Prescribing in the Elderly
Acronym: STOPP&START
Status: Completed | Type: Observational
Sponsor: Regione del Veneto - AULSS n. 7 Pedemontana (Other)
Collaborators: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Luca Pellizzari, Specialist in Geriatrics, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: 571CESC
Record Dates: First submitted 2024-11-13; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Prescriptions; Elderly (people Aged 65 or More); Hospitalized; Prevalence
Keywords: polypharmacotherapy; medication review; Drug interactions; elderly patients; deprescribin; STOPP/START criteria; of potentially inappropriate prescriptions (PIPs); potential omitted prescriptions (PPOs); PIPs; POPs; Hospital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- STOPP/START Team: Patients over 70 years old admitted to a geriatric ward, regardless of ethnicity, gender, or type of illness, will be considered eligible for enrollment. Patients transferred from another ward or admitted on a support basis to another ward will also be considered eligible.

SUMMARY:
The management of pharmacotherapy in elderly patients is an increasingly critical aspect, as polypharmacy, combined with the pharmacokinetic and pharmacodynamic changes typical of aging, makes older adults more sensitive to the development of adverse reactions. This highlights the importance of appropriate use of pharmacotherapy that considers the risks and benefits of individual treatments. The aim of this study is to measure the prevalence of pharmacological appropriateness using the STOPP/START criteria (version 2) at admission and discharge from an acute geriatric ward, thereby evaluating the impact of hospitalization on medication prescribing.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 70 years admitted to a geriatric ward
* Regardless of ethnicity, gender, or type of illness
* Patients transferred from another ward
* Patients admitted to another ward for support

Exclusion Criteria:

• Patients in the terminal phase (<6 months life expectancy)

Criteria for exit from the study (Dropout):

* Patients transferred to another hospital ward
* Patients who have deceased

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged ≥ 70 years admitted to a geriatric ward, regardless of ethnicity, gender, or type of illness, will also be considered eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of inappropriate prescribing in elderly patients at admission to an acute care hospital using STOPP/START criteria | Data collected at time Day 0 is analyzed by day 4. Data collected at time Day 1 is analyzed by day 4
  The analysis of inappropriate prescriptions at admission "Day 0" will be evaluated as a single outcome measure by aggregating data using the STOPP/START criteria. Specific assessments will be reported separately, as they involve different types of information and units of measure:
  * Prevalence of inappropriate prescriptions: The proportion of patients with prescriptions deviating from STOPP/START criteria (%).
  * Characteristics of patient history: Data such as active and passive diseases (count), place of origin (categorical variable), reason for admission (categorical variable), and presence of ADL support (binary variable: Yes/No).
  * Clinical indicators: Charlson Comorbidity Index (numerical score), number of medications (count), presence of geriatric syndromes (binary variable: Yes/No).
  * Mobility status: Whether the patient is bedridden or ambulatory (categorical variable).
  * Hospitalization history: Number of admissions in the past year (count).

SECONDARY OUTCOMES:
Prevalence of inappropriate prescribing in elderly patients at discharge from an acute care hospital using STOPP/START criteria. | Data collected at time Day 0 is analyzed by day 4. Data collected at time Day 1 is analyzed by day 4
  This analysis focuses on the prevalence of inappropriate prescriptions at discharge "Day 1", defined according to adherence to or deviation from the recommendations specified in the STOPP/START criteria.
  -Prevalence of Inappropriate Prescriptions (%): The proportion of patients with prescriptions deviating from the STOPP/START criteria.
  -Destination After Discharge: Categorical variable (e.g., home alone, home with assistance, nursing home, rehabilitation unit).
  * Length of Stay (Days)
  * Presence of Geriatric Syndromes (delirium, cognitive decline, urinary ) during Hospitalization Unit of Measurement: Binary variable (Yes/No).
  * Barthel Index at Discharge Unit of Measurement: Numerical score (in points). Description: The Barthel Index score at the time of discharge. Information for each outcome measure will be obtained from discharge letters and from the physician who cared for the patient for the majority of the hospitalization.
Percentage of cases in which inappropriate prescribing will be detected at admission and discharge | Data collected at time Day 0 is analyzed by day 4. Data collected at time Day 1 is analyzed by day 4
  Percentage of cases in which inappropriate prescriptions are identified at the time of admission "Day 0" and discharge "Day 1" for each of the individual STOPP/START criteria, i.e., for each of its recommendations.
Association between the prevalence of inappropriate prescriptions and clinical variables, measured using univariate and multivariate regression. | Data collected at time Day 0 is analyzed by day 4. Data collected at time Day 1 is analyzed by day 4
  The association between the prevalence of inappropriate prescriptions at the time of admission "Day 0" and discharge "Day 1" and clinical variables of interest (such as place of origin, level of care, comorbidities, polypharmacy, and multidimensional geriatric assessment) was analyzed using univariate and multivariate regression. The univariate regression explored the association of each variable with the prevalence of inappropriate prescriptions, while the multivariate regression was used to estimate the simultaneous effect of multiple variables, controlling for potential confounding factors.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Pellizzari Dr. Pellizzari, DR, Principal Investigator — Regione del Veneto - AULSS n. 7 Pedemontana
Locations (1):
- Regione del Veneto - AULSS n. 7 Pedemontana, Santorso, Vicenza, Italy

IPD SHARING:
Plan to Share IPD: No
IPD must be submitted to local Ethical Committee